CLINICAL TRIAL: NCT03423784
Title: Performance and Tolerability of a New Medical Device Coating Gel for the Temporary Relief of Teething Symptoms: a Randomized, Open Label, Parallel-group, Multicentre Study
Brief Title: Performance and Tolerability of a New Medical Device Gel, a Randomized, Open Label, Parallel-group, Multicentre Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BPX11-13
Record Dates: First submitted 2018-01-26; First posted 2018-02-06 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Tooth Disease
Keywords: teething in infants and children; oral gels; paediatric dentistry
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HA BPX V3.3 (Experimental): A HMWHA gel available in a formulation specificaly designed for use in infants
  Interventions: Device: HA BPX V3.3
- Dentinox-Gel N (Active Comparator): Gold standard for teething symptoms
  Interventions: Other: Dentinox-Gel N

INTERVENTIONS:
Device: HA BPX V3.3 — medical device containing HA
  Arms: HA BPX V3.3
Other: Dentinox-Gel N — Anaesthetic gel
  Arms: Dentinox-Gel N

SUMMARY:
Medical device study for efficacy and tolerability of a HA gel in the management of teething symptoms

DETAILED DESCRIPTION:
Due to the potential toxicity that can result from the use of topical anesthetics to relieve the symptoms associated with gingival inflammatory conditions or gums trauma in infant, recently, products containing Hyaluronic Acid (HA) have been marketed in Europe. In particular, Bioplax Limited is developing several high molecular weight HA medical devices characterized by the absence of preservatives, alcohol and dyes; therefore, the administration of these products in infants is safe and can help creating a natural protective layer on the gingival tissue. In previous clinical trials with these high molecular weight HA medical devices it was noted a periodontal tissue/fluid balance with accelerated healing and repair properties that could be of interest either for accelerating the wound healing process or for treating the complex physical symptoms (i.e. soreness and swelling of gums, crying, sleeplessness) related to the teething in infants. These data were confirmed by a recent pilot study on 18 infants suffering by teething where the two formulation of the tested high molecular weight HA medical device evidenced, at the end of treatment period, a statistically significant reduction of pain, swelling, gingival rush, hyper-salivation and redness, from baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female infants aged between 3 and 36 months.
2. Teething diagnosed by the presence of at least 3 of the following clinical symptoms:

   * pain
   * swelling
   * hyper-salivation
   * redness
   * abnormal teeth depth.
3. At the moment of inclusion no subcutaneous mucosal laceration must be yet appeared.
4. Infants and parents who are in a general position to follow all study requirements.
5. Informed consent form signed by parents or legal representative.

Exclusion Criteria:

1. Infants in hospitalization and/or immobilization and/or confinement to bed.
2. Infants with known history of severe renal insufficiency and/or known history of severe cardiac dysfunction and/or liver problems.
3. Use of topical oral Lidocaine, other topical oral anesthetic products and/or topical Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) within one day before inclusion.
4. Use of systemic NSAIDs within 3 days before inclusion and/or use of systemic anesthetics within 10 days before.
5. Concomitant use during the period of study of NSAIDs and/or any other anesthetics (except Dentinox®-Gel N, for subjects allocated to group II of treatment).
6. Subjects with known family history of allergic or adverse reactions to drugs or substances.
7. Infants whose parents suffer from any form of psychiatric disorder or other condition which, in the opinion of the Investigator, might invalidate the required prescription and/or observation or complicate communication with the subject.
8. Infants simultaneously participating or having participated in the last month before Visit 1 in another clinical trial.

Ages: 3 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2013-11-15 (Actual); Primary Completion 2015-03-31 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
changes in gingival swelling | 3 days
  Face, Legs, Activity, Cry and Consolability Pain Assesment Scale

SECONDARY OUTCOMES:
changes in crying | 7 days
  Face, Legs, Activity, Cry and Consolability Pain Assesment Scale

CONTACTS AND LOCATIONS:
Overall Officials: Rosu Serban, MD, Principal Investigator — SCM Dr. ROSU

IPD SHARING:
Plan to Share IPD: No